CLINICAL TRIAL: NCT05813119
Title: Comparison of Efficacy in Diagnosing of Middle Ear Pathology Between Digital Otoscope and Otoendoscope.
Brief Title: Efficacy of Digital Otoscope and Otoendoscope for Diagnosis of Middle Ear Pathology
Acronym: otoscopy
Status: Completed | Type: Observational
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Suwicha Isaradisaikul Kaewsiri, Principal Investigator, Chiang Mai University
Other Study IDs: ENT-2564-08562
Record Dates: First submitted 2022-07-31; First posted 2023-04-14 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Middle Ear Disease; Diagnosis
Keywords: Middle Ear Disease; otoscope; Diagnosis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For diagnosis of external and middle ear diseases, an otoscope is a key instrument to use. A microscope has been used as a reference standard to confirm pathology. An endoscope has been also widely used. Both microscope and endoscope provide an excellent image quality, can record and capture the images, and the images can be visualized with an export system.

A digital otoscope is widely available and more affordable. A comparative study of the efficacy of the endoscope and the digital endoscope will be performed.

DETAILED DESCRIPTION:
A comparative study for the diagnosis of middle ear disease usingTeslong digital otoscope, model MS450D39, and the otoendoscope will be performed. The participants will be recruited at the ENT clinic, University Hospital. A handheld otoscope will be used to identify the patients who have the pathology of the middle ear.

The images will be captured with both endoscopes and will be reviewed by staff, residents training in ENT, and residents training in ENT and family medicine.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with middle ear disease after examination by conventional otoscope at ENT clinic, Chiang Mai University Hospital
* Had otoscopic examination with both digital otoscope and otoendoscope in the same visit in one ear or both ears

Exclusion Criteria:

* Having abnormal external ear canals such as external auditory canal stenosis, otitis external, otomycosis, or pus/ debris in the ear canal that obscures the view of the eardrum
* Changing the pathology of the ear canal or middle ear in the same visit
* Trauma after otoscopic examination
* can not record or focus the entire view of the eardrum by both otoscopes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visit at ENT clinic, Chiang Mai University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
efficacy of digital otoscope and otoendoscope in diagnosis of middle ear pathology | 6 months
  agreement percentage
efficacy of digital otoscope and otoendoscope in diagnosis of middle ear pathology | 6 months
  Cohen's kappa coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Suwicha K Isaradisaikul, MD, Principal Investigator — Department of Otolaryngology , Faculty of Medicine, Chiang Mai University
Locations (1):
- Department of Otolaryngology Faculty of Medicine, Chiang Mai University 110 Intawaroros Road, Sriphum, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rappaport KM, McCracken CC, Beniflah J, Little WK, Fletcher DA, Lam WA, Shane AL. Assessment of a Smartphone Otoscope Device for the Diagnosis and Management of Otitis Media. Clin Pediatr (Phila). 2016 Aug;55(9):800-10. doi: 10.1177/0009922815593909. Epub 2015 Jul 7. No abstract available. PMID 26156976
- [Result] Moshtaghi O, Sahyouni R, Haidar YM, Huang M, Moshtaghi A, Ghavami Y, Lin HW, Djalilian HR. Smartphone-Enabled Otoscopy in Neurotology/Otology. Otolaryngol Head Neck Surg. 2017 Mar;156(3):554-558. doi: 10.1177/0194599816687740. Epub 2017 Jan 24. PMID 28118550
- [Result] Bhavana K, Ahmad M, Sharma P. Smartphone Otoscopy Sans Attachment: A Paradigm Shift in Diagnosing Ear Pathologies. OTO Open. 2018 Jul 19;2(3):2473974X18786496. doi: 10.1177/2473974X18786496. eCollection 2018 Jul-Sep. PMID 31565683
- [Result] Mousseau S, Lapointe A, Gravel J. Diagnosing acute otitis media using a smartphone otoscope; a randomized controlled trial. Am J Emerg Med. 2018 Oct;36(10):1796-1801. doi: 10.1016/j.ajem.2018.01.093. Epub 2018 Jan 31. PMID 29544905
- [Result] Chan KN, Silverstein A, Bryan LN, McCracken CE, Little WK, Shane AL. Comparison of a Smartphone Otoscope and Conventional Otoscope in the Diagnosis and Management of Acute Otitis Media. Clin Pediatr (Phila). 2019 Mar;58(3):302-306. doi: 10.1177/0009922818812480. Epub 2018 Nov 21. PMID 30463434